CLINICAL TRIAL: NCT00747162
Title: Correlation Between Muscle Oxygenation and Skin Pigmentation
Brief Title: Muscle Oxygenation and Skin Pigmentation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: incorporated into other study
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thomas Moore, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00009004
Record Dates: First submitted 2008-08-27; First posted 2008-09-04 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Muscle Oxygenation; Skin Pigmentation
Keywords: Compartment Syndrome; Muscle Oxygenation; Skin Pigmentation
MeSH Terms: conditions — Pigmentation Disorders; Compartment Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): We will use The INVOS cerebral oximeter to determine oxygen content in the healthy muscle. In addition, we will use a the DermaSpectrometer to determine if there are differences in our readings according to skin color.
  Interventions: Device: Measure of muscle oxygenation; Device: Skin pigmentation determination

INTERVENTIONS:
Device: Measure of muscle oxygenation — The investigators will use an INVOS oxymeter for muscle oxygenation measure.
Device: Skin pigmentation determination — The investigators will use a DermaSpectrometer to get a reading from subjects' skin color

SUMMARY:
The investigators plan to enroll 500 consecutive Subjects at a major trauma center for this study. For each patient, the body mass index (BMI), age, sex, diastolic pressure and mean arterial pressure (MAP) at time of measurements. Additional information including diseases such as diabetes and vascular disorders will be recorded. Social demographics including alcohol and tobacco use will be recorded. This is important as alcohol and tobacco use could also contribute to cardiovascular diseases. The skin pigmentation of each subject will be recorded. Two different methods will be used for this measurement. Each patient will be graded on a six point scale as described by Young (Young, 1997). Additionally, each subject will have their skin measured using a reflectance colorimeter. The colorimeter, DermaSpectrometer II (cyberDerm, Broomall, PA) uses visible light to measure the amount of light reflected off the skin. By measuring the light reflectance, the skin pigmentation can be measure (Clarys, 2000). Muscle oxygenation will be measured using a continuous dual wavelength near infrared spectrometer. Using the different absorption characteristics of deoxyhemoglobin and oxyhemoglobin, the concentration of oxyhemoglobin in the muscle at an approximate depth of 2.5 cm is determined. The INVOS cerebral oximeter (Somanetics, Troy, MI) will be used for all measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between the ages of 18 and 75 years old
* Subjects that have no lower extremity injuries.
* Subject who are classified as being either light or dark skin pigmentation.
* Subjects willing to participate in the study.

Exclusion Criteria:

* Patients with previous injury to either lower extremity
* Patients with previously diagnosed vascular disease or insufficiency
* Patients with pulmonary insufficiency or severe pulmonary injury
* Patients not willing to consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Measure from The INVOS cerebral oximeter and DermaSpectrometer | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J. Moore, MD, Principal Investigator — Emory University, Department of Orthopaedics
Locations (1):
- Grady Healthcare System, Atlanta, Georgia, United States